CLINICAL TRIAL: NCT04785495
Title: Prevalence of Anticipatory Nausea and Vomiting in Cancer Patients Exposed to Highly Emetogenic Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto Brasileiro de Controle do Cancer (Other)
Responsible Party: Principal Investigator, Rafaela de Brito Alves, Principal Investigator, Instituto Brasileiro de Controle do Cancer
Other Study IDs: 32148820000000072
Record Dates: First submitted 2021-03-01; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2020-12

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: Nausea; Antiemetics; Antineoplastic; Quality of Life
MeSH Terms: conditions — Vomiting; Nausea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer Patients Exposed to Highly Emetogenic Chemotherapy: Patients who will start chemotherapy with a high-grade emetogenic scheme and who have received adequate antiemetic prophylaxis.
  Interventions: Other: Quality-of-life assessment

INTERVENTIONS:
Other: Quality-of-life assessment — Patients will be provided the Functional Living Index - Emesis (FLIE) quality of life survey to be completed at time zero (before the application of chemotherapy) and then after 6 day, after application of chemotherapy.

SUMMARY:
Chemotherapy induced nausea and vomiting are common adverse events related to oncologic treatments. It can have deleterious effect on patients' quality of life and could lead to dose reductions and/or discontinuation of treatment. This study aims to quantify the prevalence of nausea and vomiting induced by highly emetogenic chemotherapy in patients who had adequate antiemetic prophylaxis, also to describe the epidemiologic profile and identify predisposing factors.

DETAILED DESCRIPTION:
The investigators will track patients in the first and second cycles of chemotherapy. Information regarding comorbidities, medical history and sociodemographic characteristics will be collected. The impact of nausea and vomiting induced by the treatment on patient's quality of life will be evaluated using the questionnaire Functional Living Index-Emesis - FLIE.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological confirmation of cancer;
* Patients who will start chemotherapy with a high-grade emetogenic scheme and who have received adequate antiemetic prophylaxis;
* No previous cancer treatment for the current diagnosis (excluding surgery);

Exclusion Criteria:

* Patients who have an inability to answer the questionnaire, due to lack of discernment to answer the questions reliably;
* Patients who report vomiting during the 24 hours prior to the first cycle of chemotherapy treatment;
* Patients who have a disease or condition that could cause emesis (ie, metastasis in the central nervous system, gastrointestinal obstruction or metabolic and electrolyte imbalances);
* Patients using opioids or illicit drugs;
* Alcoholism;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is estimated to recruit a sample of 50 cancer patients, undergoing chemotherapy with high emetogenic grade regimens, at the reference hospital in São Paulo, Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Prevalence of anticipatory nausea and vomiting in cancer patients undergoing highly emetogenic chemotherapy regimen | Baseline to 6 days after chemotherapy
  The prevalence of nausea and vomiting will be determined by the percentage of patients reporting the presence of a symptom at the assessment time point. Participants are asked to report any episodes of nausea and vomiting before (baseline) and up to 6 days after receiving chemotherapy. This result is measured during the first and second cycles of chemotherapy for each patient.

SECONDARY OUTCOMES:
Patient's daily diary | At the end of Cycle 1 up to the day of Cycle 2 (each cycle is 15 to 21 days)
  Participants must record any episodes of nausea and vomiting in the diary. In addition, the patient must present a score for his symptom, from zero to ten (0 = no symptom / 10 = strong symptom) using the Visual Numerical Analog Scale.
Quality of life - Functional Living Index-Emesis (FLIE) | Days 1 (before starting chemotherapy) and 6 (after chemotherapy)
  The FLIE questionnaire will be completed on days 1 (before starting chemotherapy) and 6 (after chemotherapy). The FLIE questionnaire consists of a nausea domain and a vomiting domain of nine items each where the patient should rate how much nausea and vomiting have affected the quality of life. For each question the patient will rate how much nausea (or vomiting) has affected an aspect of his quality of life during the past five days. Each question uses a visual analogue scale (where 1= no emesis-7=a great deal).

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Vieira de Rebouças, MD, Study Chair — Instituto Brasileiro de Controle do Cancer; Louize Caroline Marques Oliveira, MD, Study Chair — Instituto Brasileiro de Controle do Cancer; Rafaela de Brito Alves, MD, Principal Investigator — Instituto Brasileiro de Controle do Cancer
Locations (1):
- Rafaela de Brito Alves, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No